CLINICAL TRIAL: NCT06114173
Title: Efficacy and Safety Study of Cardunolizumab in Soft Tissue Sarcoma After Failure of at Least Anthracycline-based Chemotherapy: a Single-arm Clinical Trial
Brief Title: Efficacy and Safety Study of Cardunilizumab in Soft Tissue Sarcoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202303215
Record Dates: First submitted 2023-10-06; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-09

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- drug-dosing group (Experimental): Cardunolizumab 6mg/kg was administered every 2 weeks, with the first evaluation at 8 weeks of treatment and subsequent evaluations every 12 weeks.
  Interventions: Drug: Cardunilizumab

INTERVENTIONS:
Drug: Cardunilizumab — Cardunolizumab 6mg/kg was administered every 2 weeks, with the first evaluation at 8 weeks of treatment and subsequent evaluations every 12 weeks.
  Other Names: PD-1/CTLA-4 Bispecific Antibody

SUMMARY:
The goal of this type of study: clinical trial is to observe the efficacy and safety of cardunilizumab in soft tissue sarcomas after failure of at least first-line anthracycline-based chemotherapeutic agents, including undifferentiated sarcoma (UPS), smooth muscle sarcoma, mucinous fibrosarcoma, and poorly differentiated/undifferentiated/polymorphic liposarcoma, etc.) . The main question[s] it aims to answer are:

* Cardunilizumab is effective in soft tissue sarcomas after failure of at least first-line anthracycline-based chemotherapeutic agents, including undifferentiated sarcoma (UPS),smooth muscle sarcoma, mucinous fibrosarcoma, and poorly differentiated/undifferentiated/polymorphic liposarcoma) is effective .
* Cardunilizumab has manageable adverse effects. Participants will be given Cardunolizumab 6mg/kg once every 2 weeks free

DETAILED DESCRIPTION:
Some important factors for applying for this clinical trial:

1. sarcomas are dangerous, subtypically complex, and lack effective treatment. Soft Tissue Sarcoma treatment is looking for new drugs to improve patient prognosis.
2. PD-1 inhibitor monotherapy has shown initial efficacy in some soft tissue sarcoma subtypes.
3. Dual immunotherapy targeting PD-1 and CTLA-4 is more effective in the treatment of malignant tumors.
4. The "two-in-one" dual-antibody cardunculizumab, which is more potent and less toxic, has been approved for marketing by the Fast Track Review.
5. We hypothesize that the treatment of soft tissue sarcoma with cadunilizumab is safer and more effective than currently available immunotherapy options; however, this has not yet been reported.

ELIGIBILITY:
Inclusion Criteria:

1. agree to sign the informed consent form.
2. 18 years ≤ age < 75 years.
3. Pathologic subtypes include undifferentiated sarcoma (UPS), smooth muscle sarcoma, mucinous fibrosarcoma, poorly differentiated/ dedifferentiated/ pleomorphic Liposarcoma; diagnosis confirmed by pathology at a tertiary care hospital.
4. soft tissue sarcoma evaluated as metastatic or inoperable.
5. previous systemic therapy including at least anthracycline-based chemotherapeutic agents.
6. at least one measurable lesion (CT or MRI); Tissue specimen which can be safely obtained by vacutainer before and during treatment.
7. ECOG physical status score of 0-1.
8. an expected survival time of >12 weeks.
9. Normal major organ function, i.e., the following criteria are met:

   a) Hematology: i. Absolute neutrophil count ANC ≥ 1.5 × 109/L (1,500/mm3). ii. Platelet count ≥ 80 × 109/L (80,000/mm3 ). iii.Hemoglobin ≥ 90 g/L. b) Liver: i. Serum total bilirubin (TBil) ≤ 1.5 × ULN. ii. AST and ALT ≤ 2.5 × ULN. iii. serum albumin (ALB) ≥ 28 g/L. iv. serum bilirubin (ALB) ≤ 1.5 × ULN. c) Coagulation function: i. International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN.

   d) Cardiac function: i. Left ventricular ejection fraction (LVEF) ≥ 50%.
10. Female subjects of childbearing potential must undergo a urine or serum pregnancy test within 3 days prior to the first dose (if the urine pregnancy test is not confirmed).
11. The subject is willing and able to comply with the schedule of visits, treatment regimens, laboratory tests, and other requirements of the study.

Exclusion Criteria:

1. patients with active (symptomatic) brain metastases; or uncontrolled medical conditions with severe insufficiency of vital organ function including liver, kidney, heart, lung or bone marrow.
2. subjects with active viral hepatitis B, inactive or asymptomatic hepatitis B virus (HBV) carriers with HBV DNA greater than 1000 IU/mL; and subjects with active viral hepatitis C.
3. a history of known positive tests for human immunodeficiency virus or known acquired immunodeficiency syndrome.
4. active or potentially relapsing autoimmune disease;
5. history of severe allergic reaction to any monoclonal antibody and/or components of the study drug.
6. known active tuberculosis TB and subjects suspected of having active TB will be required to undergo a clinical examination to exclude known active syphilis infection.
7. history of non-infectious pneumonia/interstitial lung disease requiring systemic glucocorticoid therapy or current non-infectious pneumonia.
8. a serious infection occurring within 4 weeks prior to the first dose, including, but not limited to, an active infection with comorbidities requiring hospitalization, sepsis, or severe pneumonia treated with systemic anti-infective therapy within 2 weeks prior to the first dose.
9. serious illness or concomitant non-neoplastic conditions such as neurological disorders, psychiatric disorders, infectious diseases, or laboratory abnormalities.
10. major surgical procedure or serious traumatic injury within 30 days prior to the first dose of the drug, or major surgical procedure planned within 30 days of the first dose of the drug; minor localized surgical procedures within 3 days prior to the first dose of the drug
11. known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
12. subjects requiring systemic therapy with corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive drugs within 14 days prior to administration of study drug. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted. Topical, ocular, intra-articular, intranasal and inhaled corticosteroids are permitted in subjects. Physiologic replacement doses of systemic corticosteroids are allowed, even if >10 mg/day of prednisone equivalent. Short-term use of corticosteroids for prevention or treatment of non-autoimmune diseases is permitted.
13. Patients with clinically significant cardiovascular disease; 1) Myocardial infarction, unstable angina, pulmonary embolism, aortic coarctation, deep vein thrombosis, and any arterial thromboembolic event within 6 months prior to dosing; 2) New York Heart Association (NYHA) heart failure ≥ Class II; 3) Severe arrhythmias requiring long-term pharmacologic intervention; asymptomatic atrial fibrillation with stable ventricular rate is permitted. patients; 4) Cerebrovascular event (CVA) within 6 months prior to randomization; 5) Left ventricular ejection fraction (LVEF) < 50%; 6) previous history of myocarditis or cardiomyopathy. 14.
14. concurrent enrollment in another clinical study, unless it is an observational, non-interventional clinical study or an interventional study.
15. currently undergoing treatment for cancer (chemotherapy, radiotherapy, immunotherapy, or biologic therapy).
16. prior treatment with anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody.
17. have received a live vaccine within 30 days prior to the first dose or plan to receive a live vaccine during the study period.
18. known history of mental illness, substance abuse, alcoholism, or drug addiction.
19. pregnant or breastfeeding female.
20. any pre-existing or current medical condition, treatment, or laboratory test abnormality that could confound the results of the study, interfere with the subject's ability to participate in the study throughout the study, or participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate，ORR | 24 months
  Tumor volume reduction of up to 30%（According to RECIST 1.1 efficacy evaluation criteria）

SECONDARY OUTCOMES:
Incidence of adverse events | 24 months
  according to criteria CTCAE 5.0,the ratio of AE and SAE which were defined by the common terminology criteria for adverse events,CTCAE.
Incidence of immune-related adverse events | 24 months
  Adverse effects due to the use of immunotherapy
overall survival,OS | 24 months
  Time from initiation of immunotherapy to death or time lost to visit.
progression-free survival,PFS | 24 months
  Time from initiation of immunotherapy to disease progression or death from other causes.

OTHER OUTCOMES:
PD-L1 immunohistochemical assay values | 24MONTHS
  Immunohistochemical testing values for all patients were completed by our pathology department

CONTACTS AND LOCATIONS:
Overall Officials: bin Li, doctor, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
we will share the some dates to the website:http://www.medresman.org.cn/login.aspx or publication of results of clinical trials in the form of papers

REFERENCES:
- [Result] Savina M, Le Cesne A, Blay JY, Ray-Coquard I, Mir O, Toulmonde M, Cousin S, Terrier P, Ranchere-Vince D, Meeus P, Stoeckle E, Honore C, Sargos P, Sunyach MP, Le Pechoux C, Giraud A, Bellera C, Le Loarer F, Italiano A. Patterns of care and outcomes of patients with METAstatic soft tissue SARComa in a real-life setting: the METASARC observational study. BMC Med. 2017 Apr 10;15(1):78. doi: 10.1186/s12916-017-0831-7. PMID 28391775
- [Result] Tawbi HA, Burgess M, Bolejack V, Van Tine BA, Schuetze SM, Hu J, D'Angelo S, Attia S, Riedel RF, Priebat DA, Movva S, Davis LE, Okuno SH, Reed DR, Crowley J, Butterfield LH, Salazar R, Rodriguez-Canales J, Lazar AJ, Wistuba II, Baker LH, Maki RG, Reinke D, Patel S. Pembrolizumab in advanced soft-tissue sarcoma and bone sarcoma (SARC028): a multicentre, two-cohort, single-arm, open-label, phase 2 trial. Lancet Oncol. 2017 Nov;18(11):1493-1501. doi: 10.1016/S1470-2045(17)30624-1. Epub 2017 Oct 4. PMID 28988646